CLINICAL TRIAL: NCT02743338
Title: CompRest - a Randomized Comparison Between Sleep Compression and Sleep Restriction for the Treatment of Insomnia
Brief Title: CompRest - a Comparison Between Sleep Compression and Sleep Restriction for Treating Insomnia
Acronym: CompRest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Research Group Leader, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/44-31/4
Record Dates: First submitted 2016-04-12; First posted 2016-04-19 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Insomnia
Keywords: Sleep Restriction; Sleep Compression; Cognitive Behavioral Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sleep Restriction followed by additional CBT-i components (Experimental): Sleep Restriction treatment during 5+5 weeks. Followed by being offered an additional intervention consisting of other ICBT-i components during 10 weeks.
  Interventions: Behavioral: Sleep Restriction; Behavioral: Additional CBT-i components
- Sleep Compression followed by additional CBT-i components (Active Comparator): Sleep Compression treatment during 5+5 weeks. Followed by being offered an additional intervention consisting of other ICBT-i components during 10 weeks.
  Interventions: Behavioral: Sleep Compression; Behavioral: Additional CBT-i components
- Sleep Restriction followed by no intervention (Active Comparator): Sleep Restriction treatment during 5+5 weeks. Followed by NOT being offered or informed of an additional intervention consisting of other ICBT-i components during 10 weeks.
  Interventions: Behavioral: Sleep Restriction
- Sleep Compression followed by no intervention (Active Comparator): Sleep Compression treatment during 5+5 weeks. Followed by NOT being offered or informed of an additional intervention consisting of other ICBT-i components during 10 weeks.
  Interventions: Behavioral: Sleep Compression

INTERVENTIONS:
Behavioral: Sleep Restriction — Behavioral component of CBT-i. Sleep restrictions includes curtailing bed time to match sleep time as registered during the first week of treatment, and expanding bed time contingent upon increased sleep efficiency, until optimal balance between sleep time and sleep efficiency is reached. The first five weeks, therapist support is provided via written messages. The next five weeks, patient works independently. At the end of tenth treatment week, therapist and patient make plan for future.
  Arms: Sleep Restriction followed by additional CBT-i components; Sleep Restriction followed by no intervention
Behavioral: Sleep Compression — Behavioral component of CBT-i. Sleep compression includes gradually compressing bed time over several weeks to approach sleep time as registered during the first week of treatment, and stopping compression when optimal balance between sleep time and sleep efficiency is reached. The first five weeks, therapist support is provided via written messages. The next five weeks, patient works independently. At the end of tenth treatment week, therapist and patient make plan for future.
  Arms: Sleep Compression followed by additional CBT-i components; Sleep Compression followed by no intervention
Behavioral: Additional CBT-i components — After 5+5 weeks of either Sleep Restriction or Sleep Compression, a randomized sample from each treatment Group is offered additional components of CBT-i, such as Stimulus Control, Cognitive Restructuring, Relaxation and Visualization for 10 weeks, without therapist support. Component allocation based on individual analysis.
  Arms: Sleep Compression followed by additional CBT-i components; Sleep Restriction followed by additional CBT-i components

SUMMARY:
This study includes two consecutive sub-trials.

Cognitive Behavioral Therapy (CBT) is treatment of choice for Insomnia. One of the most important treatment Components in CBT for insomnia (CBT-i) is Sleep Restriction (SR), but lately, adverse effects related to SR have been reported. A treatment method with similarities to SR is Sleep Compression (SC). SC is not as well studied as SR, but appears to have similar effects to SR but without the adverse effects. The first sub-trial thus aims at directly comparing SR and SC. The second sub-trial aims at evaluating any additional effects of CBT-i components given as an add-on treatment to a randomized selection of half participants in each original treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia Disorder according to DSM-V
* Sufficient language skills
* Having access to Internet to fill out forms and participating in treatment
* Not foresee obstacles to participating in treatment during the coming 20 weeks, or participating in measurements during the coming year.

Exclusion Criteria:

* Sleep disorders requiring other treatment
* High consumption of alcohol/drugs that affect sleep
* Somatic or psychiatric conditions counter-indicative of treatments given in the study, requiring acute care, or with symptoms and level of functioning affecting the ability to participate in the treatment programs.
* Working (night) shifts
* Ongoing psychological treatment for Insomnia with sleep restriction or sleep compression as a treatment component - also previous such treatment can be excluding
* Use of sleep medication in such a way that may hinder the implementation of the methods in this treatment
* Pre-treatment measurements not finished within the given time-frame.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from base-line to 5 weeks, 10 weeks, 20 weeks and 57 weeks
  7-item, self-rated questionnaire measuring change in insomnia severity. Bastien, C. H., Vallières, A., & Morin, C. M. (2001). Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Medicine, 2, 297-307.

SECONDARY OUTCOMES:
Sleep diary | Continuously from one week before treatment start (-1 week) to the last week of treatment (week 10)
  Daily self-ratings on a number of sleep parameters, resulting in measures of sleep latency, total sleep time, sleep efficacy, number of nighttime awakenings, subjective sleep quality and daytime functioning
Actigraphy | Continuously from one week before treatment start (-1 week) to the last week of treatment (week 10)
  An actigraph is placed on the participant's arm for one week. They measure participants' activity in the form of movements. It will be used for acquiring sleep data and calculate sleep latency, total sleep time, sleep efficacy, number of nighttime awakenings and daytime activity
Adverse Events | Week 2, week 4 and week 5
  Self-report questionnaires and interviews
Sleep Problems Acceptance Questionnaire | Change from base-line to 5 weeks, 10 weeks, 20 weeks and 57 weeks

OTHER OUTCOMES:
Polysomnography | One week before treatment (Week -1) and at week 1, week 3, week 5, and week 10
  Ambulatory objective sleep stage and sleep timing measure

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienheten (Internet Psychiatry Clinic) Psykiatri Sydväst, SLSO, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jernelov S, Rosen A, Forsell E, Blom K, Ivanova E, Maurex L, Jansson-Frojmark M, Akerstedt T, Kaldo V. Is sleep compression therapy non-inferior to sleep restriction therapy? A single-blind randomized controlled non-inferiority trial comparing sleep compression therapy to sleep restriction therapy as treatment for insomnia. Sleep. 2025 Aug 14;48(8):zsaf093. doi: 10.1093/sleep/zsaf093. PMID 40205789
- [Derived] Kraepelien M, Blom K, Forsell E, Hentati Isacsson N, Bjurner P, Morin CM, Jernelov S, Kaldo V. A very brief self-report scale for measuring insomnia severity using two items from the Insomnia Severity Index - development and validation in a clinical population. Sleep Med. 2021 May;81:365-374. doi: 10.1016/j.sleep.2021.03.003. Epub 2021 Mar 16. PMID 33813233